CLINICAL TRIAL: NCT06799208
Title: Evaluating the Efficacy of Laparoscopic Approach in Adhesive Intestinal Obstruction
Brief Title: Laparoscopic Approach in Adhesive Intestinal Obstruction
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Sayed Mohammad Ibrahim, DR, Assiut University
Other Study IDs: Laparoscopic adhesiolysis
Record Dates: First submitted 2025-01-10; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Efficacy of Laparoscopic Adhesiolysis
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patient diagnosed with intestinal obstruction
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Minimal invasive approach. Have peritoneal tissue sparing character . Minimal blood loss . Reduction of postoperative adhesions.

SUMMARY:
A Clinical trail to evaluate the efficacy of Laparoscopic approach in Adhesive Intestinal Obstruction .

DETAILED DESCRIPTION:
There was a rapid growth of minimally invasive operations. Through its peritoneal tissue sparing character and minimal blood loss, laparoscopy was soon claimed to reduce adhesion formation and associated complications.

The aim of this prospective clinical trial study is to evaluate the use of laparoscopy in management of clinically diagnosed adhesive intestinal obstruction and the criteria of selection to get the best results .

ELIGIBILITY:
Inclusion Criteria:

* Patient who clinically diagnosed as adhesive intestinal obstruction.
* Both sexes
* Adult patients (above 18 years old

Exclusion Criteria:

* • Patient refused to participate in this study.

  * Patients not fit for laparoscopic surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to General Surgery department with adhesive intestinal obstruction during the year of study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of days post- operative till passing stool . | 1 year

IPD SHARING:
Plan to Share IPD: No